CLINICAL TRIAL: NCT06156423
Title: Investigation of the Effect of Motor Control Exercises Given With Telerehabilitation on Shoulder Function and Quality of Life in Patients Undergoing Rotator Cuff Surgery
Brief Title: Investigation of the Effect of Motor Control Exercises in Patients Undergoing Rotator Cuff Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sinem Yenil, PT, PhD, Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-390737
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2023-12

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff surgery; telerehabilitation; motor control
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Control Rehabilitation (Experimental)
  Interventions: Other: Motor control exercise
- Standard Rehabilitation (Active Comparator)
  Interventions: Other: Standard exercise

INTERVENTIONS:
Other: Motor control exercise — Motor control exercises include stabilization exercises for the scapula with external focus by activating the correct alignment and kinetic chain by providing verbal feedback and visual feedback.
  Arms: Motor Control Rehabilitation
Other: Standard exercise — The standard rehabilitation group received a rehabilitation program via video call 3 days a week for 12 weeks.
  Arms: Standard Rehabilitation

SUMMARY:
The aim of the study is to examine the effect of motor control exercises given through telerehabilitation on shoulder function and quality of life in patients undergoing rotator cuff surgery.

DETAILED DESCRIPTION:
Treatment of rotator cuff tears can be conservative or surgical. The aim of rehabilitation postoperative period, is to reduce pain, increase joint range of motion (ROM), and enable the patient to return to normal functional activities as soon as possible while preventing the repaired tissue from tearing again.

Motor control training based on motor control theory reorganizes the cerebral cortex. In people with shoulder pain, a scapulothoracic posture retraining program reduces shoulder pain and improves scapulothoracic movement and muscle activation patterns and shoulder function. Therefore, rehabilitation should include correct positioning of the scapulothoracic joint through active muscle activation (motor control training) and retraining. However, the evidence is still limited and the effect of motor control exercises is not yet fully understood. Over the last 15 years, telerehabilitation in the broader field of telehealth has been used to help patients in rural areas improve healthcare and access services to reduce cost and transportation issues. Studies on the upper extremity have also begun to increase in recent years. The aim of the study is to examine the effect of motor control exercises given through telerehabilitation on shoulder function and quality of life in patients undergoing rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergone rotator cuff surgery
* being 18 years of age
* agree to participate in the study,
* allowed early rehabilitation after surgery,
* can speak and understand Turkish
* can make video conferences and phone calls.

Exclusion Criteria:

* have had previous surgery on the affected shoulder,
* have neurological deficits and motor control disorders,
* have systemic rheumatological disease,
* have developed any complications that may affect rehabilitation in the shoulder,
* have had revision surgery on the affected shoulder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Pain assessment will be evaluated with the Visual Analog Scale (VAS) before surgery, at the 6th week and at the 12th week after surgery, during activity, rest and sleep. As the score increases, it indicates that the pain increases.
Shoulder Range of Motion Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Range of motion of the shoulder will be evaluated with a electrogoniometer. Evaluations will be made actively for shoulder flexion, abduction, internal and external rotation and active total elevation
Active Internal Rotation Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  In active internal rotation of the shoulder, the distance between the thumb and the T5 spinous process will be measured with a tape measure.
Scapular Dyskinesis Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Scapular dyskinesis will be evaluated with the lateral scapular glide test.
Shoulder muscle strength assessment | Preoperative and postoperative 12th week
  Shoulder abduction, flexion, internal and external rotation and scaption muscle strength will be measured with a dynamometer.
Grip strength assessment | Preoperative and postoperative 12th week
  Grip strength will be evaluated with a Jamar hand dynamometer.
Shoulder function assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Shoulder function will be evaluated with Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. The total score is 100, with higher scores indicating more disability.
Shoulder function assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Other shoulder function assessment will be evaluated with American Shoulder and Elbow Surgeons Scale (ASES). A combination of these scores will yield an ASES score ranging from 0 (absence of function) to 100 (normal function).
Kinesiophobia Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Kinesiophobia assessment will be evaluated with Tampa Scale of Kinesiophobia. The total score varies between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia.
Sleep quality assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Sleep quality will be evaluated with Pittsburgh Sleep Quality Index (PSQI). The overall score ranges from 0 to 21. Lower scores indicate better sleep quality.
Quality of Life Assessment | Preoperative, postoperative 6th week and postoperative 12th week
  Quality of life will be evaluated with the Western Ontario Rotator Cuff Index (WORC), specific to rotator cuff injuries. The total score ranges from 0 to 2100, with lower scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinem Yenil, Denizli, Denizli, Turkey (Türkiye)